CLINICAL TRIAL: NCT01904292
Title: A Phase Ib, Open-Label, Multicenter Study to Investigate the Pharmacokinetics, Pharmacodynamics, and Safety of Tocilizumab Following Subcutaneous Administration to Patients With Systemic Juvenile Idiopathic Arthritis
Brief Title: A Study of Subcutaneously Administered Tocilizumab in Participants With Systemic Juvenile Idiopathic Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA28118; 2012-003490-26 (EudraCT Number)
Record Dates: First submitted 2013-06-14; First posted 2013-07-22 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

ARMS (1):
- Tocilizumab (Experimental): Participants will receive SC dose of tocilizumab based on body weight; participants with <30 kg will receive 162 milligrams (mg) of tocilizumab Q2W and those participants =>30 kg will receive 162 mg of tocilizumab QW, for 52 weeks.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Subcutaneous 162 mg dose QW or Q2W for 52 weeks
  Other Names: RoActemra/Actemra

SUMMARY:
This open-label, multicenter study will evaluate the pharmacokinetics, pharmacodynamics, and safety of subcutaneously administered tocilizumab in participants with Systemic Juvenile Idiopathic Arthritis (sJIA). Participants with body weight less than (<) 30 kilograms (kg) will receive subcutaneous (SC) tocilizumab dose every 2 weeks (Q2W) and participants with body weight greater than or equal to (>=) 30 kg will receive weekly (QW), for 52 weeks. Tocilizumab was administered every 10 days until pre-planned interim analysis was performed and changed to Q2W in participants with body weight <30 kg.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sJIA according to the International League of Associations for Rheumatology (ILAR) classification
* History of inadequate clinical response (in the opinion of the treating physician) to Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) and corticosteroids
* If a participant has received previous treatment with any biologic agents other than tocilizumab, these must have been discontinued according to the timelines defined by protocol prior to the baseline visit
* Participants currently receiving tocilizumab by the intravenous (IV) route of administration and with well-controlled disease do not require a period of discontinuation of IV tocilizumab and should have their first dose of SC tocilizumab administered on the date that their next IV tocilizumab infusion would be due
* Concurrent treatment with Disease Modifying Anti-Rheumatic Drugs (DMARDs) including methotrexate (MTX), NSAIDs, and oral corticosteroids are permitted at the discretion of the investigator
* Participants of reproductive potential must be willing to use highly effective contraceptive methods

Exclusion Criteria:

* Prior discontinuation of IV tocilizumab because of inadequate clinical response or safety events (including hypersensitivity)
* Participants with poorly controlled disease (in the opinion of the treating physician) despite current treatment with IV tocilizumab
* sJIA that is well controlled by any treatment agent other than tocilizumab (Juvenile Arthritis Disease Activity Score of 71 Joints [JADAS-71] less than or equal to [<=] 3.8 with no fever)
* Participants who are wheelchair-bound or bedridden
* Any other auto-immune, rheumatic disease, or overlapping syndrome other than sJIA
* Lack of recovery from recent surgery or an interval of <6 weeks since surgery at the time of the screening visit
* Females who are pregnant, lactating, or intending to become pregnant during study conduct
* Any significant concurrent medical or surgical condition that would jeopardize the participant's safety or ability to complete the study
* Known Human Immunodeficiency Virus (HIV) infection or other acquired forms of immune compromise or inborn conditions characterized by a compromised immune system
* History of alcohol, drug, or chemical abuse within 6 months of screening
* Any active acute, subacute, chronic, or recurrent bacterial, viral, or systemic fungal infection or any major episode of infection requiring hospitalization or treatment during screening or treatment with IV antibiotics completed within 4 weeks of the screening visit or oral antibiotics completed within 2 weeks of the screening visit
* History of atypical tuberculosis (TB) or active TB requiring treatment within 2 years prior to screening visit
* Positive TB test at screening unless treated with anti-TB therapy for at least 4 weeks prior to receiving study drug
* History of reactivation or new onset of a systemic infection such as herpes zoster or Epstein-Barr virus within 2 months of the screening visit
* Hepatitis B surface antigen or hepatitis C antibody positivity or chronic viral or autoimmune hepatitis
* History of concurrent serious gastrointestinal disorders such as ulcer or inflammatory bowel disease, Crohn's disease, ulcerative colitis, or other symptomatic lower gastrointestinal conditions
* History of or current cancer or lymphoma
* Uncontrolled diabetes mellitus with elevated glycosylated hemoglobin
* Macrophage activation syndrome (MAS) within 3 months of the screening visit
* Inadequate hematologic, renal or liver function

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2013-08-15 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of Tocilizumab | Age <2 years: 0 hours(h) on Days(D) 0,84; on D5,14,42,70,85,88,98,182,266, 364. Weight <30kg, Age>=2 years: 0,6,12h on D0,84; on D2,5,14,42,56,70,86,87,88,90,98,182,266,364. Weight >=30kg: 0,6,12h on D0, 91; on D2,4,7,14,28,56,92,93,95,96,98,182,266, 364
Pharmacokinetics: Maximum Plasma Concentration (Cmax) of Tocilizumab | Age <2 years: 0h on D0,84; on D5,14,42,70,85,88,98,182,266,364. Weight <30 kg, Age >=2 years: 0,6,12h on D0,84; on D2,5,14,42,56,70,86,87,88,90,98,182,266,364. Weight >=30 kg: 0,6,12h on D0, 91; on D2,4,7,14,28,56,92,93,95,96,98,182,266,364
Pharmacokinetics: Minimum Plasma Concentration (Cmin) of Tocilizumab | Weight <30 kg: predose (0h) on Days 0 and 84. Weight >= 30 kg: predose (0h) on Days 0 and 91

SECONDARY OUTCOMES:
Pharmacodynamics: Serum Interleukin-6 (IL6) Levels | Age<2 years: 0h on Days 0,84; Days 5,14,42,70,85,88,98,182,266,364. Weight <30 kg, Age >=2 years: 0,6,12h on Days 0,84; Days 2,5,14,42,56,70,86,87,88,90,98,182,266,364. Weight >=30kg: 0,6,12h on Days 0,91;Days 2,4,7,14,28,56,92,93,95,96,98,182,266,364
Pharmacodynamics: Soluble IL-6 Receptor (sIL-6R) Levels | Age<2 years: 0h on Days 0,84; Days 5,14,42,70,85,88,98,182,266,364. Weight <30 kg, Age >=2 years: 0,6,12h on Days 0,84; Days 2,5,14,42,56,70,86,87,88,90,98,182,266,364. Weight >=30kg: 0,6,12h on Days 0,91;Days 2,4,7,14,28,56,92,93,95,96,98,182,266,364
Pharmacodynamics: Serum C-Reactive Protein (CRP) Levels | Age <2years: Days 0,14,28,42,70,84,98,126, 154,182,210,238,266,294,322,350,364. Weight <30 kg, Age >=2years: Days 0,14,28,42,70, 98,126,154,182,210,238,266,294,322,350,364. Weight >=30kg: Days 0,7,14,21,28,42, 56,70,84,91,95,96,98,182,266,294,322,350,364
Pharmacodynamics: Serum Erythrocyte Sedimentation Rate (ESR) | Age <2years: Days 0,14,28,42,70,84,98,126, 154,182,210,238,266,294,322,350,364. Weight <30 kg, Age >=2years: Days 0,14,28,42,70, 98,126,154,182,210,238,266,294,322,350,364. Weight >=30kg: Days 0,7,14,21,28,42, 56,70,84,91,95,96,98,182,266,294,322,350,364
Pharmacodynamics: Percentage of Participants with Anti-Tocilizumab Antibodies | Age <2 years: Days 0, 84, 182, 266, 364. Weight <30 kg, Age >=2 years: Days 0, 84, 182, 266, 364. Weight >=30 kg: Days 0, 91, 182, 266, 364
Safety: Percentage of Participants with At Least 1 Adverse Event | 57 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (42):
- United States (11):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Connecticut Children's Medical Center; 5E Clinical Trials Unit, Hartford, Connecticut
  - Ann & Robert H. Lurie Children's Hospital of Chicago; Division of Rheumatology, Chicago, Illinois
  - The University of Chicago;Department of Pediatrics, Chicago, Illinois
  - Hackensack University Medical Center; Pediatric Rheumatology, Hackensack, New Jersey
  - Levine Children's Hospital; Divison of Pediatric Rheumatology; Department of Pediatrics, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children'S Hospital Medical Center; Division of Rheumatology, Cincinnati, Ohio
  - Cleveland Clinic Fndn, Cleveland, Ohio
  - University of Utah; Immunology/Rheumatology/Allergy, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Argentina (2):
  - Hospital Gral de Niños Pedro Elizalde, Buenos Aires
  - Hospital de Ninos de la Santisima Trinidad; Reumatologia Infantil, Córdoba
- Australia (2):
  - Westmead Hospital; Paediatric Rheumatology, Westmead, New South Wales
  - Royal Children'S Hospital; Paediatric Rheumatology, Parkville, Victoria
- Brazil (3):
  - Hospital das Clinicas - FMUSP Ribeirao Preto; Pediatria - Imunologia e Reumatologia, Ribeirão Preto, São Paulo
  - Hospital das Clinicas - FMUSP; Instituto da Crianca - Reumatologia, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESP, São Paulo, São Paulo
- Canada (3):
  - Alberta Children'S Hospital, Calgary, Alberta
  - Children'S Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital For Sick Children, Toronto, Ontario
- CH de Bicêtre; Pediatrie Generale, Le Kremlin-Bicêtre, France
- Germany (3):
  - Charité Campus; Virchow Klinikum Berlin, Berlin
  - Uniklinikum Freiburg Zentrum für Kinder- und Jugendmedizin; Pädiatrische Infektio- u. Rheumatologie, Freiburg im Breisgau
  - Asklepios Klinik; Zentrum fuer Allgemeine Paediatrie und Neonatologie, Sankt Augustin
- Italy (3):
  - Irccs Ospedale Pediatrico Bambin Gesu - Dip. Di Medicina, Rome, Lazio
  - Istituto Giannina Gaslini-Ospedale Pediatrico IRCCS, Genoa, Liguria
  - Nuovo Ospedale Pediatrico Meyer; Reumatologia - Clinica Pediatrica 1°, Florence, Tuscany
- Mexico (3):
  - Hospital Infantil de México "Federico Gomez"; Rheumatology, México
  - Cliditer SA de CV, Miexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez; Pediatria, Monterrey
- Russia (2):
  - FSBI "Scientific Research Institute of Rheumatology" of russian Academy of Medical Sciences, Moscow
  - SI Sceintific children health center RAMS, Moscow
- Spain (5):
  - Hospital Sant Joan De Deu; Servicio de Reumatologia Pediatrica, Esplugas de Llobregat, Barcelona
  - Hospital Infantil Universitario Niño Jesus, Servicio Reumatologia, Madrid
  - Hospital Ramon y Cajal ; Servicio de Reumatologia, Madrid
  - Hospital de La Paz; Unidad de Reumatologia Pediatrica, Madrid
  - Hospital Universitario la Fe: Servicio de Reumatologia Pediatrica, Valencia
- United Kingdom (4):
  - Bristol Royal Hospital For Children, Bristol
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital; Somers Clinical Research Facility, London
  - Nottingham Children's Hospital, Nottingham

REFERENCES:
- [Derived] Ruperto N, Brunner HI, Ramanan AV, Horneff G, Cuttica R, Henrickson M, Anton J, Boteanu AL, Penades IC, Minden K, Schmeling H, Hufnagel M, Weiss JE, Pardeo M, Nanda K, Roth J, Rubio-Perez N, Hsu JC, Wimalasundera S, Wells C, Bharucha K, Douglass W, Bao M, Mallalieu NL, Martini A, Lovell D, Benedetti F; Paediatric Rheumatology INternational Trials Organisation (PRINTO) and the Paediatric Rheumatology Collaborative Study Group (PRCSG). Subcutaneous dosing regimens of tocilizumab in children with systemic or polyarticular juvenile idiopathic arthritis. Rheumatology (Oxford). 2021 Oct 2;60(10):4568-4580. doi: 10.1093/rheumatology/keab047. PMID 33506875